CLINICAL TRIAL: NCT01292525
Title: Prospective, Multicenter, Randomized, Double-blind, Controlled Parallel Group Study Designed to Assess the Risk-benefit Balance of the Gradual Withdrawal of a Calcineurin Inhibitor (Tacrolimus) in Renal Transplant Patients Over 4 Years and Clinically Selected
Brief Title: Protocol Calcineurin Inhibitor (CNI) Weaning
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Difficulties of recruitment
Sponsor: Nantes University Hospital (Other)
Responsible Party: Pr Magali GIRAL, Nantes University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 09/7-D; 2010-019574-33 (EudraCT Number)
Record Dates: First submitted 2011-02-08; First posted 2011-02-09 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2015-05

CONDITIONS: Function of Renal Transplant
Keywords: Withdrawal of Tacrolimus and renal graft; renal allograft; stable renal function
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tacrolimus (Active Comparator)
  Interventions: Drug: Tacrolimus
- Withdrawal of Tacrolimus (Experimental)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tacrolimus — A control group continued conventional therapy, Tacrolimus (Prograf®) ("control" group) and will be followed in parallel group "withdrawal" that will stop treatment with Tacrolimus (Prograf®).
  Arms: Tacrolimus
Drug: Placebo — Patients randomized to the "withdrawal"group will begin the protocol with their usual dose of Tacrolimus (Prograf®) (initial dose). The initial dose of tacrolimus (Prograf®) will be reduced by one third at visit 3 (day 0) and again a third visit 5 (J60). The complete withdrawal Tacrolimus (Prograf®) begins to visit 7 (J120). The withdrawal of Tacrolimus (Prograf®) will be obtained in four months. Monitoring of all patients lasted 17 months in total from the screening visit, which corresponds to 12 months after complete withdrawal of Tacrolimus (Prograf®) for patients in the "withdrawal" group.
  Arms: Withdrawal of Tacrolimus

SUMMARY:
The main objective of this study is to demonstrate the benefit of the withdrawal of Tacrolimus (Prograf®) on renal function in patients one year after the end of the weaning period. The secondary objectives will focus on assessing the risks and consequences of withdrawal of Tacrolimus (Prograf®).

ELIGIBILITY:
Pre-inclusion criteria :

* Male or female aged between 18 and 80 years (inclusive),
* Having received a deceased donor transplant or living with ABO compatibility,
* First renal allograft for at least 4 years and under 10 years,
* Presenting a stable renal function : serum creatinine with a variation of ± 25% of the average of the year before inclusion,
* Treated with tacrolimus (Prograf®) in combination with MPA (Cellcept® and Myfortic®) + / - steroids (between 5 and 10 mg per day),
* Patient has given informed consent,
* Patient insured,
* Patient (of childbearing age) with effective contraception.

Inclusion Criteria:

* Glomerular Filtration Rate (GFR), defined by the dosage of cystatin C ≥ 40 ml/min/1, 73m²,
* Proteinuria ≤ 0,5 g / day,
* Patient with serum levels of Tacrolimus between 5 to 10 ng / ml on average during the last 6 months (inclusive). It is accepted that 25% of the assays performed during the last 6 months, serum levels of tacrolimus are outside the limits mentioned above (5-10 ng / ml). They must nevertheless be between 3.5 to 12.5 ng / ml (inclusive).
* Patient with serum levels of MPA (Cellcept® and Myfortic®) higher ≥ 30 mg / ml,
* No anti-HLA antibodies at the time of inclusion, verified using highly sensitive techniques (Luminex HD),
* Lack of histological evidence of cellular or humoral acute or chronic or subclinical rejection on renal graft according to the latest classification of Banff 2009.

Exclusion Criteria:

* Patients under age 18 or over 80 years,
* Transplanted from less than 4 years and over 10 years,
* Patients re-transplanted,
* Transplantation of several organs,
* Patient not treated with tacrolimus as maintenance therapy,
* Serum levels of Tacrolimus patient <5 or >10 ng / ml,
* Serum levels of MPA of the patient <30 mg / ml,
* Patients treated with other immunosuppressive drugs that Tacrolimus (Prograf®), MPA (Cellcept® and Myfortic®) and steroids,
* Patient not having a stable graft function at baseline (change in serum creatinine > 25% of the average of the year before inclusion in the study), with a GFR defined by the dosage of cystatin C <40 ml/min/1, 73m² at the time of inclusion,- Patients with proteinuria > 0.5 g at study entry,
* Patient with HLA antibodies at study entry,
* Patient non-compliant,
* Presence of histological evidence of cellular or humoral acute or chronic or subclinical rejection on renal graft according to the latest classification of Banff 2009,
* History of lymphoproliferative disorders,
* Diagnosis of a malignancy within 5 years before enrollment,
* Significantly abnormal hematologic data of a clinical standpoint, as determined by the investigator for hematocrit, hemoglobin, white blood cell count or platelets,
* Data significantly abnormal blood biochemistry of a clinical standpoint, as determined by the investigator,
* Abuse of significant drug or alcohol at the time of inclusion, determined by the investigator,
* Patient positive for antibodies to hepatitis C or hepatitis B surface antigen of hepatitis B (HBsAg) or HIV infection,
* Participation in a clinical study within 3 months,
* Pregnancy, Breastfeeding.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-05; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Renal function | one year after complete withdrawal of Tacrolimus
  The primary endpoint will be the improvement of renal function one year after complete withdrawal of Tacrolimus (Prograf®) assessed by measuring the glomerular filtration rate (GFR) calculated by the dosage of cystatin C according to the equation Bricon. The DFG will be compared between times J-30 and J480 (1 year after the withdrawal).

SECONDARY OUTCOMES:
Renal function | one year after complete withdrawal
  Improvement of renal function by measuring serum creatinine, using the original MDRD equation,
Acute rejection | one year after complete withdrawal
  Rate of histologically proven acute rejection by biopsy according to Banff classification 2009,
Chronic rejection | One year after complete withdrawal
  Rate of chronic rejection histologically proven by biopsy according to Banff classification 2009,
Steroid-resistant rejection | One year after complete withdrawal
  Rates of steroid-resistant rejection
Graft survival | One year after complete withdrawal
  Rate of return to dialysis (graft survival)
Cancer and infections | one year after complete withdrawal
  Incidence of cancer and infections
Patients survival | One year after complete withdrawal
  Survival rate of patients
Anti-HLA antibodies | One year after complete withdrawal
  Appearance of anti-HLA donor specific and non-donor specific antibodies measured by the technique Luminex
Histological lesions of rejection | One year after complete withdrawal
  The appearance of histological lesions of cellular or humoral acute or chronic or subclinical rejection on the biopsy protocol
Histological lesions of fibrosis | One year after complete withdrawal
  Onset or worsening of histological lesions of interstitial fibrosis and tubular atrophy on biopsy inflammatory
Hypertension, hyperglycemia and hyperlipidemia | One year after complete withdrawal
  Incidence of hypertension, hyperglycemia and hyperlipidemia
Quality of life | One year after complete withdrawal
  Determination of the benefits of withdrawal of Tacrolimus on the quality of life of patients, defined by the scale of quality of life validated SF-36 used at the beginning (J-15) and at the end of the weaning period (J120) at 6 months (J300) and one year after complete withdrawal of Tacrolimus (J480)

CONTACTS AND LOCATIONS:
Overall Officials: Magali GIRAL, Profesor, Principal Investigator — Nantes University Hospital; Jean-Paul SOULILLOU, Profesor, Study Chair — Nantes University Hospital; Christophe LEGENDRE, Profesor, Study Chair — Hôpital Necker - AP-HP; Emmanuel MORELON, Profesor, Study Chair — Hospices Civils de Lyon; Georges MOURAD, Profesor, Study Chair — CHU de Montpellier
Locations (1):
- Nantes University Hospital, Nantes, France

REFERENCES:
- [Derived] Masset C, Dantal J, Soulillou JP, Walencik A, Delbos F, Brouard S, Giral M; Nantes DIVAT Consortium. Case Report: Long-term observations from the tacrolimus weaning randomized clinical trial depicts the challenging aspects for determination of low-immunological risk patients. Front Immunol. 2022 Nov 28;13:1021481. doi: 10.3389/fimmu.2022.1021481. eCollection 2022. PMID 36518770